CLINICAL TRIAL: NCT04731168
Title: Prevention of Sleep Apnea After General Anaesthesia With a Mandibular Advancement Device: a Randomized Controlled Trial
Brief Title: Prevention of Sleep Apnea After General Anaesthesia With a MAD
Acronym: PoMAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, Program director of regional anaesthesia, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-01177
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Peri-operative Medicine; Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Occlusal Splints

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- MAD (Experimental): Patients will have a mandibular advancement device during the first postoperative night
  Interventions: Device: Mandibular advancement device

INTERVENTIONS:
Device: Mandibular advancement device — Patients will have a mandibular advancement device during the first postoperative night
  Arms: MAD

SUMMARY:
Sleep apneic episodes increase after general anaesthesia up to the third postoperative night. A mandibular advancement device, called MAD, is a small device that is inserted in the patient's mouth during the night and allows the advancement of the mandible, preventing sleep apneic episodes. The objective of this randomized controlled trial is to determine whether a MAD reduces the impact of general anaesthesia on the increase of the sleep apneic episodes in the postoperative period. All patients will have their sleep-related respiratory data measured using a portable respiratory polygraphy recorder (ResMed Embletta® system). This portable recorder allows a non-invasive recording of nasal airflow through a nasal cannula, oxygen saturation (SpO2) via finger pulse oximetry, respiratory efforts through thoracic and abdominal belts, and body position.

ELIGIBILITY:
Inclusion Criteria:

- adult patient undergoing any lower limb surgery

Exclusion Criteria:

* continuous positive airway pressure (CPAP) treatment for obstructive sleep apnoea,
* presence of severe respiratory or cardiovascular disease
* preoperative consumption of benzodiazepine,
* chronic use of opioids > 30 mg/day morphine equivalent
* no tooth
* patient known for malignant hyperthermia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Supine AHI | Postoperative night 1
  Apnea-Hypopnea index in the supine position

SECONDARY OUTCOMES:
Global AHI | Postoperative night 1
  Gobal Apnea-Hypopnea index: the number of apnoea and hypopnoea per hour of recording
OAI | Postoperative night 1
  Obstructive apnoea index: the number of apnoea from an obstructive origin per hour of recording
CAI | Postoperative night 1
  Central apnoea index: the number of apnoea from a central origin per hour of recording
Hypopnea index | Postoperative night 1
  Hypopnea index: the number of hypopnoea per hour of recording
ODI | Postoperative night 1
  Obstruction desaturation index: number of oxygen desaturation (≥3%) episodes per hour of sleep.
Respiratory Rate | Postoperative night 1
  Respiratory Rate
Percentage of supine time | Postoperative night 1
  Percentage of supine time

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois and University of Lausanne, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided